CLINICAL TRIAL: NCT03160079
Title: A Phase I/II Study of Blinatumomab in Combination With Pembrolizumab (MK-3475) for Adults With Relapsed or Refractory B-lineage Acute Lymphoblastic Leukemia With High Bone Marrow Lymphoblast Percentage
Brief Title: Blinatumomab & Pembrolizumab for Adults With Relapsed/Refractory B-cell ALL With High Marrow Lymphoblasts
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Amgen (Industry)
Responsible Party: Principal Investigator, James Mangan, Associate Clinical Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161287/UCHMC1504
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: B-Cell Acute Lymphoblastic Leukemia, Adult
Keywords: blinatumomab; pembrolizumab; MK-3475; relapsed; refractory; B-lineage acute lymphoblastic leukemia; ALL
MeSH Terms: conditions — Burkitt Lymphoma; Recurrence | interventions — blinatumomab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blinatumomab + Pembrolizumab (Experimental): Drug: blinatumomab Cycle 1 Blinatumomab Day 1-7 Continuous IV infusion for 28 days (9 mcg/day) Blinatumomab Day 8-28 Continuous IV infusion for 28 days (28 mcg/day)
  Cycle 2-5 Blinatumomab Day 1-28 Continuous IV infusion for 28 days (28 mcg/day)
  Cycle length 42 days
  Other Names:
  Blincyto
  Drug: pembrolizumab Cycle 1 Pembrolizumab Day 15 and 36 IV infusion over 30 minutes (200mg)
  Cycle 2-5 Pembrolizumab Day 15 and 36 IV infusion over 30 minutes (200mg)
  Other Names:
  * Keytruda
  * MK-3475
  Interventions: Drug: blinatumomab; Drug: pembrolizumab

INTERVENTIONS:
Drug: blinatumomab — Cycle 1 Blinatumomab Day 1-7 Continuous IV infusion for 28 days (9 mcg/day) Blinatumomab Day 8-28 Continuous IV infusion for 28 days (28 mcg/day)
  Cycle 2-5 Blinatumomab Day 1-28 Continuous IV infusion for 28 days (28 mcg/day)
  Cycle length 42 days
  Other Names: Blincyto
Drug: pembrolizumab — Cycle 1 Pembrolizumab Day 15 and 36 IV infusion over 30 minutes (200mg)
  Cycle 2-5 Pembrolizumab Day 15 and 36 IV infusion over 30 minutes (200mg)
  Other Names: Keytruda; MK-3475

SUMMARY:
This is a Phase I/II study of blinatumomab in combination with pembrolizumab in adult patients with relapsed or refractory B-lineage ALL (B-ALL). The primary objective of this study is to determine if the addition of pembrolizumab to blinatumomab improves the Complete Response Rate (CR) and Complete Remission with Partial Hematologic Recovery (CRh) relative to blinatumomab alone in adult subjects with relapsed or refractory B-cell acute lymphoblastic leukemia with high bone marrow lymphoblast percentage (>50% lymphoblasts).

DETAILED DESCRIPTION:
This is a Phase I/II study of blinatumomab in combination with pembrolizumab in adult patients with relapsed or refractory B-lineage ALL (B-ALL). The primary objective of this study is to determine if the addition of pembrolizumab to blinatumomab improves the Complete Response Rate (CR) and Complete Remission with Partial Hematologic Recovery (CRh) relative to blinatumomab alone in adult subjects with relapsed or refractory B-cell acute lymphoblastic leukemia with high bone marrow lymphoblast percentage (>50% lymphoblasts).

Mechanisms of resistance to blinatumomab are not well understood although inhibition of or suboptimal T-cell activation may play an important role. Programmed Death-Ligand 1 (PD-L1) and Programmed Death-Ligand 2 (PD-L2) expression and upregulation in lymphoblasts and the bone marrow microenvironment at baseline and in response to cytokines including those released upon blinatumomab exposure may inhibit T-cell function through the Programmed Death 1 (PD-1) receptor and lead to resistance to blinatumomab. The investigators hypothesize that part of the resistance to therapy with blinatumomab is mediated by the exuberant cytokine release seen with higher disease burden leading to increased expression of PD-L1 and PD-L2. Enhancing T-cell activity through use of the PD-1 inhibitor pembrolizumab is predicted to augment the activity of blinatumomab and convert more patients to complete remission and prolong remission durations. This study will also act to expand knowledge of PD-L1 and PD-L2 dynamics in response to blinatumomab. It will also be a paradigm for the addition of checkpoint inhibitors to therapy with bifunctional T-cell engaging antibodies currently in development for targeting other liquid and solid tumors.

The PD-1 receptor-ligand interaction is a major pathway hijacked by tumors to suppress immune control. This suggests that the PD-1/PD-L1 pathway plays a critical role in tumor immune evasion and should be considered as an attractive target for therapeutic intervention. Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the Immunoglobulin G4 (IgG4/kappa) isotype designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.

The study will be conducted in 2 stages:

Stage 1 is to ensure safety of pembrolizumab in combination with blinatumomab.

Stage 2 of the study will include an expansion cohort of up to 21 additional subjects (for a total of 24 subjects) to evaluate the efficacy of the combination of blinatumomab and pembrolizumab in adults with relapsed/refractory B-cell ALL

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory B-lineage acute lymphoblastic leukemia (B-ALL) having received at least 1 prior line of therapy
* Philadelphia chromosome positive (Ph+), or Breakpoint Cluster Region Protein-Abelson Murine Leukemia Viral Oncogene Homolog 1 (BCR-ABL1) positive B-lineage ALL must have failed at least 1 second or third generation tyrosine kinase inhibitor (TKI) or be intolerant to TKIs
* Greater than 50% lymphoblasts on screening bone marrow aspirate or biopsy
* Adequate organ function
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.
* A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Male subjects must agree to use a latex condom during sexual contact with females of childbearing potential even if they have had a successful vasectomy starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Allogeneic hematopoietic cell transplantation within 5 years of study drug administration
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) or Granulocyte Colony-Stimulating Factor (G-CSF) use within 2 weeks of study treatment and throughout the study
* Prior checkpoint inhibitor therapy including anti Programmed Death Receptor 1 (anti-PD1), anti-PD-L1, anti-CTLA4 (cytotoxic T-lymphocyte-associated protein 4), anti tumor necrosis factor receptor superfamily, member 9 (anti-CD137), or anti-PD-L2 therapy
* Active Central Nervous System (CNS) or testicular involvement by leukemia
* History of neurologic disorder
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Burkitt lymphoma/leukemia
* Has a diagnosis of congenital immunodeficiency
* Has a known history of active Bacillus Tuberculosis (TB)
* Known Human Immunodeficiency Virus (HIV) infection
* Active hepatitis B or hepatitis C infection
* Has received a live vaccine within 30 days prior to first dose
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* History of autoimmune disease
* Known interstitial lung disease
* Any evidence of active, non-infectious pneumonitis or has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Patients who have received chemotherapy or radiotherapy within 2 weeks prior to entering the study or has not recovered from adverse events due to agents administered more than 2 weeks earlier.
* Patients who are less than 4 weeks from surgery or have insufficient recovery from surgical-related trauma or wound healing.
* Known impaired cardiac function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2023-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James K Mangan, M.D., P.h.D., Principal Investigator — University of California, San Diego
Locations (4):
- United States (4):
  - UCSF Fresno Community Cancer Institute, Clovis, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC Irvine Health Chao Family Comprehensive Cancer Center, Orange, California
  - UCSF Comprehensive Cancer Center, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Weber JS. Practical management of immune-related adverse events from immune checkpoint protein antibodies for the oncologist. Am Soc Clin Oncol Educ Book. 2012:174-7. doi: 10.14694/EdBook_AM.2012.32.79. PMID 24451730
- [Background] Weber JS, Kahler KC, Hauschild A. Management of immune-related adverse events and kinetics of response with ipilimumab. J Clin Oncol. 2012 Jul 20;30(21):2691-7. doi: 10.1200/JCO.2012.41.6750. Epub 2012 May 21. PMID 22614989
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Weber J, Thompson JA, Hamid O, Minor D, Amin A, Ron I, Ridolfi R, Assi H, Maraveyas A, Berman D, Siegel J, O'Day SJ. A randomized, double-blind, placebo-controlled, phase II study comparing the tolerability and efficacy of ipilimumab administered with or without prophylactic budesonide in patients with unresectable stage III or IV melanoma. Clin Cancer Res. 2009 Sep 1;15(17):5591-8. doi: 10.1158/1078-0432.CCR-09-1024. Epub 2009 Aug 11. PMID 19671877
- [Background] Lemech C, Arkenau HT. Novel treatments for metastatic cutaneous melanoma and the management of emergent toxicities. Clin Med Insights Oncol. 2012;6:53-66. doi: 10.4137/CMO.S5855. Epub 2012 Jan 5. PMID 22253555
- [Background] Phan GQ, Weber JS, Sondak VK. CTLA-4 blockade with monoclonal antibodies in patients with metastatic cancer: surgical issues. Ann Surg Oncol. 2008 Nov;15(11):3014-21. doi: 10.1245/s10434-008-0104-y. Epub 2008 Aug 21. PMID 18716842
- [Background] Bristol-Myers Squibb: YERVOY (ipilimumah): Serious and fatal immune-mediated adverse reactions--YERVOY Risk Evaluation and Mitigation Strategy (REMS). http://www.yervoy.com/hcp/rems.aspx
- [Background] Bristol-Myers Squibb: YERVOY (ipilimumab) prescribing information revised March 2011. http://www.accessdata.fda.gov/drugsatfda _ docs/label/2011/1253 77s0000lbl.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Blinatumomab + Pembrolizumab: Drug: blinatumomab Cycle 1 Blinatumomab Day 1-7 Continuous IV infusion for 28 days (9 mcg/day) Blinatumomab Day 8-28 Continuous IV infusion for 28 days (28 mcg/day)
  Cycle 2-5 Blinatumomab Day 1-28 Continuous IV infusion for 28 days (28 mcg/day)
  Cycle length 42 days
  Other Names:
  Blincyto
  Drug: pembrolizumab Cycle 1 Pembrolizumab Day 15 and 36 IV infusion over 30 minutes (200mg)
  Cycle 2-5 Pembrolizumab Day 15 and 36 IV infusion over 30 minutes (200mg)
  Other Names:
  * Keytruda
  * MK-3475
  blinatumomab: Cycle 1 Blinatumomab Day 1-7 Continuous IV infusion for 28 days (9 mcg/day) Blinatumomab Day 8-28 Continuous IV infusion for 28 days (28 mcg/day)
  Cycle 2-5 Blinatumomab Day 1-28 Continuous IV infusion for 28 days (28 mcg/day)
  Cycle length 42 days
  pembrolizumab: Cycle 1 Pembrolizumab Day 15 and 36 IV infusion over 30 minutes (200mg)
  Cycle 2-5 Pembrolizumab Day 15 and 36 IV infusion over 30 minutes (200mg)
- Blinatumomab Only: Patients did not receive Pembrolizumab due to early termination
Period: Overall Study
Arm/Group | Blinatumomab + Pembrolizumab | Blinatumomab Only
Started | 12 | 4
Completed Course 1 | 8 | 4
Completed Course 2 | 5 | 0
Completed Course 3 | 3 | 0
Completed Course 4 | 1 | 0
Completed Course 5 | 1 | 0
Completed | 8 | 4
Not Completed | 4 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Disease Progression | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographics were recorded for all patients who enrolled
Groups:
- Blinatumomab + Pembrolizumab: Drug: blinatumomab Cycle 1 Blinatumomab Day 1-7 Continuous IV infusion for 28 days (9 mcg/day) Blinatumomab Day 8-28 Continuous IV infusion for 28 days (28 mcg/day) Cycle 2-5 Blinatumomab Day 1-28 Continuous IV infusion for 28 days (28 mcg/day) Cycle length 42 days
  Other Names:
  Blincyto Drug: pembrolizumab Cycle 1 Pembrolizumab Day 15 and 36 IV infusion over 30 minutes (200mg) Cycle 2-5 Pembrolizumab Day 15 and 36 IV infusion over 30 minutes (200mg)
  Other Names:
  Keytruda MK-3475 blinatumomab: Cycle 1 Blinatumomab Day 1-7 Continuous IV infusion for 28 days (9 mcg/day) Blinatumomab Day 8-28 Continuous IV infusion for 28 days (28 mcg/day) Cycle 2-5 Blinatumomab Day 1-28 Continuous IV infusion for 28 days (28 mcg/day) Cycle length 42 days pembrolizumab: Cycle 1 Pembrolizumab Day 15 and 36 IV infusion over 30 minutes (200mg) Cycle 2-5 Pembrolizumab Day 15 and 36 IV infusion over 30 minutes (200mg)
- Total: Total of all reporting groups
Arm/Group | Blinatumomab + Pembrolizumab | Blinatumomab Only | Total
Number analyzed (Participants) | 12 | 4 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 3 | 14
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 2 | 11
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 10 | 1 | 11
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (ORR)
Description: Best overall response rate (ORR) with the combination of blinatumomab and pembrolizumab in adult subjects with relapsed or refractory B-cell acute lymphoblastic leukemia will be defined as the Complete Response (CR) rate plus the Complete Response with Hematologic Recovery (CRh) rate after treatment of combination therapy. According to the National Comprehensive Cancer Network (NCCN) Guidelines for Acute Lymphoblastic Leukemia (version 1, 2015), CR is defined as <5% lymphoblast in the bone marrow without evidence of circulating lymphoblasts or extramedullary disease. CRh is defined as for CR except with platelet count >50,000/microliter, hemoglobin >7 g/dL, and neutrophil (ANC) >500/microliter.
Time Frame: 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab + Pembrolizumab | Blinatumomab Only
Number analyzed (Participants) | 12 | 4
Participants
  Complete Response (CR) | 6 | 0
  Complete Response with Hematologic Recovery | 1 | 0
  Partial Response | 1 | 0
  Refractory | 4 | 1
  Not Evaluated | 0 | 3

2. Secondary Outcome: Complete Response Rate (CR)
Description: CR is defined as <5% lymphoblast in the bone marrow without evidence of circulating lymphoblasts or extramedullary disease.
Time Frame: 28 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Blinatumomab Only: Participants who did not receive Pembrolizumab due to early termination
Arm/Group | Blinatumomab + Pembrolizumab | Blinatumomab Only
Number analyzed (Participants) | 12 | 4
Participants | 6 | 0

3. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate in Subjects Achieving a CR or CRh
Description: Minimal residual disease (MRD) negativity in subjects achieving a CR or CRh will be defined as less than 0.01% residual lymphoblasts by multiparameter flow cytometry.
Time Frame: 28 weeks
Population: 7 participants received both Blinatumomab and Pembrolizumab and achieved a CR or CRh. Of the 7, 6 had achieved MRD negativity and 1 had unevaluable data. 2 participants received only Blinatumomab and achieved a CR or CRh, but neither had evaluable MRD data.
Measure: Count of Participants; unit: Participants
Arm/Group | Blinatumomab + Pembrolizumab | Blinatumomab Only
Number analyzed (Participants) | 7 | 2
Participants
  MRD negativity | 6 | 0
  MRD not evaluable | 1 | 2

4. Secondary Outcome: 2 Year Relapse-free Survival Rate
Description: The number of patients achieving relapse free survival at 2 years. Relapse-free survival (RFS) will be defined as the time from achieving CR or CRh to relapse defined as the reappearance of lymphoblasts in bone marrow or blood at >5% of cells or reappearance of extramedullary disease.
Time Frame: 2 years
Population: All participants who achieved a CR or CRh response were in the Blinatumomab + Pembrolizumab group. No participants in the Pembrolizumab Only group achieved a CR or CRh.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Blinatumomab + Pembrolizumab
Number analyzed (Participants) | 7
participants | 2 [1 to 7]

5. Secondary Outcome: 2-year Overall Survival Rate
Description: The number of participants achieving survival at 2 years. 2-year overall survival (OS) will be defined as the time from starting study therapy to death from any cause.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Blinatumomab + Pembrolizumab: Number of participants who received both study drugs
- Pembrolizumab Only: Number of patients who only received Pembrolizumab
Arm/Group | Blinatumomab + Pembrolizumab | Pembrolizumab Only
Number analyzed (Participants) | 12 | 4
participants | 3 [2.55 to 4.95] | 1 [.85 to 1.65]

ADVERSE EVENTS:
Time Frame: 8 months (7 months on treatment and 30 days monitoring post last dose). Note that overall survival was monitored for 2 years, but Adverse Events were not monitored after 8 months.
Description: Adverse events were collected via regular investigator assessments and regular laboratory testing.
Groups:
- Blinatumomab + Pembrolizumab: Patients who received both study drugs
Arm/Group | Blinatumomab + Pembrolizumab | Blinatumomab Only
All-Cause Mortality (participants affected / at risk) | 1/12 | 0/4
Serious Adverse Events (participants affected / at risk) | 4/12 | 1/4
Other Adverse Events (participants affected / at risk) | 12/12 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinatumomab + Pembrolizumab (N=12) | Blinatumomab Only (N=4)
Cytokine Release Syndrome (Immune system disorders) | 1 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute Disseminating Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Macrophage Activation Syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Intracranial Hemorrhage/Hematoma (Nervous system disorders) | 1 (2) | 1 (1)
Neck Edema (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinatumomab + Pembrolizumab (N=12) | Blinatumomab Only (N=4)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Alanine aminotransaminase increased (Investigations) | 4 (5) | 1 (1)
Alkaline Phosphatase Increase (Investigations) | 3 (4) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (14) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (7) | 0 (0)
Aspartate Aminotransaminase Increased (Investigations) | 4 (6) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Blood Bilirubin Increased (Investigations) | 3 (4) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Chills (General disorders) | 5 (5) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 7 (14) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Edema Limbs (General disorders) | 1 (42) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Facial Flushing (Vascular disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 5 (5) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Fever (General disorders) | 6 (14) | 2 (2)
Fluid Volume Overload (Endocrine disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 9 (11) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (3) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (11) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 5 (6) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (5) | 0 (0)
Leukocystosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — A disorder characterized by laboratory test results that indicate an increased number of white blood cells in the blood.
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) — A disorder presence of macules (flat) and papules (elevated). Also known as morbilliform rash, one of the most common cutaneous adverse events, frequently affecting the upper trunk, spreading centripetally, associated with pruritis.
Nausea (Gastrointestinal disorders) | 3 (9) | 0 (0) — A disorder characterized by a queasy sensation and/or the urge to vomit.
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — A disorder characterized by marked discomfort sensation in the neck area.
NEUTROPHIL COUNT DECREASED (Investigations) | 10 (10) | 0 (0) — A finding based on laboratory test results that indicate a decrease in number of neutrophils in a blood specimen.
PLATELET COUNT DECREASED (Investigations) | 2 (14) | 0 (0) — A finding based on laboratory test results that indicate a decrease in number of platelets in a blood specimen.
Salivary duct inflammation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — A disorder characterized by inflammation of the salivary duct.
Brachial plexopathy (Nervous system disorders) | 0 (0) | 1 (1) — A disorder characterized by regional paresthesia of the brachial plexus, marked discomfort and muscle weakness, and limited movement in the arm or hand.
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5) — A disorder characterized by of marked discomfort in the throat
Ventricular tachycardia (Cardiac disorders) | 6 (7) | 2 (2) — A disorder characterized by a dysrhythmia with a heart rate greater than 100 beats per minute that originates distal to the bundle of His.
Vomiting (Nervous system disorders) | 3 (3) | 0 (0) — A disorder characterized by the reflexive act of ejecting the contents of the stomach through the mouth.
White blood cell decreased (Investigations) | 2 (8) | 0 (0) — A finding based on laboratory test results that indicate an decrease in number of white blood cells in a blood specimen.
Aphonia (Nervous system disorders) | 0 (0) | 1 (1) — A disorder characterized by the inability to speak. It may result from injuries to the vocal cords or may be functional (psychogenic).
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — A finding of injury of the soft tissues or bone characterized by leakage of blood into surrounding tissues.
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (2) | 1 (1) — A disorder characterized by the uncontrolled shaking movement of the whole body or individual parts.
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (2) — A disorder characterized by an abnormal increase of cerebrospinal fluid in the ventricles of the brain.
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — A disorder characterized by a dysrhythmia with a heart rate greater than 100 beats per minute that originates in the sinus node.

LIMITATIONS AND CAVEATS:
There have been several limitations for reporting these results. The original PI left University of California San Diego (UCSD) and remained the Investigational New Drug (IND) holder, but UCSD is listed as the responsible reporting party on CT.gov. The final data analysis was not received until recently because of extensive technical and logistical issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT03160079/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT03160079/ICF_002.pdf